CLINICAL TRIAL: NCT04339335
Title: Pulsed Radiofrequency of the Occipital Nerves for Chronic Headache Management.
Brief Title: Pulsed Radiofrequency in Chronic Headaches
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Associate Professor of Anaesthesiology, Attikon Hospital
Other Study IDs: AttikonH PRF STUDY
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Pulsed radiofrequency of the occipital nerves — pulsed radiofrequency of the greater and lesser occipital nerves bilaterally

SUMMARY:
Pulsed radiofrequency of the occipital nerves (greater and lesser) for primary headache management.

DETAILED DESCRIPTION:
Patients participating suffered from primary headaches (migraine, cluster, and tension headache) and occipital neuralgia were enrolled in the study. They have all received in the past the standard systemic pharmacotherapy prophylaxis for headache management (with topiramate or amitriptylline) as well as tryptanes for rescue treatment, and were scheduled for a diagnostic nerve block of the occipital nerves in cases of intractable pain. Inclusion criteria included: not adequate response to systemic pharmacotherapy, pain over crises of >4/10, occipital tenderness bilaterally or unilaterally, and days with headache of more than 10/month. Exclusion criteria were age<18 years old, pregnancy or lactation, presence of cardiac pacemaker, previous therapy with PRF, severe psychiatric disorder and patient refusal. In cases of a positive response to the diagnostic nerve block with local anesthetic, with >50% pain relief they were scheduled for pulsed radiofrequency of GON and LON bilaterally.

Primary outcome measure was the days with headache per month, before and after treatment. In addition, pain during headache crisis (with Visual Analogue Scale, VAS, 0-10), the analgesic consumption (number per month) and the quality of life (measured with EQ6D) were studied. All measurements were performed before treatment, as well as after 1, 3, 6, and 12 months. All patients completed the Brief Pain Inventory questionnaire in Greek language and signed an informed consent prior treatment. All measurements were accomplished by an independed (blinded) researcher of the pain unit. All complications and side effects were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* not adequate response to systemic pharmacotherapy
* pain over crises of >4/10
* occipital tenderness bilaterally or unilaterally,
* days with headache of more than 10/month.

Exclusion Criteria:

* age<18 years old,
* pregnancy or lactation
* presence of cardiac pacemaker
* previous therapy with PRF
* severe psychiatric disorder
* severe coagulopathy
* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients participating suffered from primary headaches (migraine, cluster, and tension headache) and occipital neuralgia were enrolled in the study. They have all received in the past the standard systemic pharmacotherapy prophylaxis for headache management (with topiramate or amitriptylline) as well as tryptanes for rescue treatment, and were scheduled for a diagnostic nerve block of the occipital nerves in cases of intractable pain.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Days with headache | 12 months
  days with headache per month

SECONDARY OUTCOMES:
pain during crisis | 12 months
  pain during crisis with Numeric Rating Scale 0-10
analgesics consumption | 12 months
  number of analgesics consumption per month
quality of life | 12 months
  quality of life by EQ5D

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece

IPD SHARING:
Plan to Share IPD: No